CLINICAL TRIAL: NCT00866021
Title: A Multicenter, Randomized, Open Label, Pilot Study to Assess the Possibility of Concomitant Treatment of HCV/HIV co Infection With Peg-interferon + Ribavirin, and Lopinavir/r as a Single Antiretroviral Agent.
Brief Title: Treatment of HIV/HCV Coinfection With Peg-IFN and Ribavirin in Patients Receiving ART Monotherapy With Lopinavir/r
Acronym: PEKARI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA-5506; 2007-003544-30 (EudraCT Number)
Record Dates: First submitted 2009-03-18; First posted 2009-03-20 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2013-03

CONDITIONS: HIV/HCV Co-infection; HIV Infections
Keywords: HIV infection; HCV infection; treatment experienced
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Lopinavir; lopinavir-ritonavir drug combination; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lopinavir/ritonavir (LPV/r) as single antiretroviral administered concomitantly with peg-interferon and ribavirin
  Interventions: Drug: Lopinavir/ritonavir
- 2 (Active Comparator): Lopinavir/ritonavir (LPV/r) with 2 NRTIs, administered concomitantly with peg-interferon and ribavirin
  Interventions: Drug: Lopinavir/ritonavir with two nucleoside analogs

INTERVENTIONS:
Drug: Lopinavir/ritonavir — NRTI sparing-regimen
  Other Names: Kaletra
  Arms: 1
Drug: Lopinavir/ritonavir with two nucleoside analogs — LPV/r plus 2NRTIs + PEG-INF + RBV
  Arms: 2

SUMMARY:
The aim of this study is to assess the efficacy of lopinavir/r in monotherapy and peg-interferon plus ribavirin for the control of both HIV and HCV infection respectively after 12 months of active treatment for HCV.

DETAILED DESCRIPTION:
Viral hepatitis, mainly when caused by the hepatitis C virus (HCV), is highly significant in the setting of infection by the human immunodeficiency virus (HIV) because high activity antiretroviral therapy (HAART) has a very favorable impact upon morbidity and mortality of this disease. HAART has achieved disease control, significantly increasing survival and improving the quality of life of subjects with HIV infection.

Spain has one of the highest prevalences of HIV-HCV co-infection because both HCV and HIV infection are strongly associated to being or having been an intravenous drug user (IDU); thus, from 61% to 69% of these subjects infected by HIV in Spain are also infected by HCV.

From 1998, standard treatment for chronic C hepatitis consists of the combination of interferon alpha and ribavirin, based on an increased efficacy versus interferon monotherapy; however, development of pegylated interferon, with a more convenient bioavailability as compared to conventional interferon alpha, has allowed for developing even more effective combined therapies and the possibility of improving response prediction based on changes in viremia within the first few weeks of treatment. However, treatment of HCV infection usually involves severe side effects, which often lead to treatment discontinuation or to the need for adjusting drug dosage, in which case treatment efficacy may decrease.

HCV+ subjects who, because of HIV co-infection, should also receive HAART, may have an increased number or increased severity of adverse reactions due to interactions occurring with drug co-administration.

Lopinavir/ritonavir (LPV/r) is a potent HIV protease inhibitor and is characterized by a very high pharmacological and genetic barrier.

Different studies (subject cohorts, uncontrolled studies) during the past years have appeared in the literature showing the efficacy of LPV/r or controlling viral replication.

Most studies were conducted with the soft gel capsule formulation of LPV/r. In this study, the new formulation of LPV/r (Kaletra) as tablets approved by the FDA and EMEA (Spain authorization 30th Oct 2006) will be used. This new formulation will provide additional benefits to this strategy that has only been studied to date with soft gel capsules.

Based on the foregoing and on the additional cost savings involved in this strategy, we think that LPV/r, as single antiretroviral agent concomitantly administered with treatment for hepatitis C virus infection may provide significant benefits because it would prevent interactions between NRTIs and ribavirin, thus being potentially able to decrease the adverse events derived from mitochondrial toxicity and minimizing the possibility of anemia. In addition, replacement of NNRTIs by LPV/r may significantly decrease CNS involvement that may be enhanced by co-administration of efavirenz and peg-interferon, or minimize the risk of hepatotoxicity caused by nevirapine.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria in the 30 days prior to study inclusion.

1. Subject consent to participate in this study after being informed of all trial aspects that may influence his/her decision, given by signing and dating the informed consent form approved by the CREC of the corresponding center.
2. Subject is at least 18 years old, is co-infected by HIV and HCV, and has been recommended treatment for HCV infection.
3. Liver biopsy confirming the presence of chronic hepatitis performed within one year of patient entry into the study.
4. Undetectable viral load (<50 cop/mL) during at least the 6 last months (confirmed). At least two viral load determinations lower than 50 cop/mL 6 months apart are required. The inclusion of patients showing one single "blip" during the pre-enrollment past 6 months is allowed. A "blip" is defined as a HIV viral load greater or equal to 50 cop/mL both preceded and followed of viral loads inferior to 50 cop/mL without changes in the antiretroviral treatment.
5. CD4 at screening should be at least or greater to 350 cells/microl
6. Subject on continued, uninterrupted antiretroviral therapy for the past 6 months with

   1. LPV/r + 2 NRTIs/NtRTIs for at least 4 weeks;
   2. 1 NNRTI + 2 NRTIs
   3. 3 NRTIs Only changes in protease inhibitor due solely to toxicity, simplification, or optimization are acceptable
7. Subject has not been treated for an active opportunistic infection within 30 days of the baseline visit.
8. Subject has a Karnofsky index >-70.
9. Throughout the study, the patient does not require and agrees not to take any of the following drugs, that are contraindicated with Kaletra: astemizole, terfenadine, midazolam, triazolam, cisapride, certain ergot derivatives (ergotamine, dihydroergotamine, ergonovine, methylergonovine), pimozide, propafenone, and flecainide. Rifampin, a potent enzyme inducer, should not be administered with the study medication due to the possibility of a significant decrease in Kaletra concentrations during concomitant administration.
10. Subject agrees not to take any medication, including over-the-counter medicines, alcohol, drugs, or herbal preparations without the knowledge and approval of the principal investigator.
11. Laboratory tests have been made in the subject in the past 30 days.
12. Hemoglobin >8.0 g/dL Absolute neutrophil count >750 cells/microL Platelet count >20.000/microL ALT or AST <5 x upper normal limit (UNL) Creatinine <1.5 x UNL
13. Triglycerides <750 mg/dL.
14. For women with childbearing potential, a negative result of a pregnancy test is available and they agree to use throughout the study at least two contraceptive methods (including a barrier one) of proven reliability in the investigator's opinion.
15. In the case of men subjects, they are agreed to use during the hepatitis C treatment with ribavirin at least two contraceptive methods (including a barrier one).

Exclusion Criteria:

Subjects will be excluded from study participation if they meet any of the following criteria:

1. Subjects in whom a switch in protease inhibitor has ever been made due to suspected or documented virological failure.
2. Subjects requiring treatment with drugs whose association with LPV/r is contraindicated based on Kaletra prescribing information..
3. Active drug addiction or psychiatric disease that may prevent protocol compliance. Use of cannabis or being on methadone treatment are excepted, provided protocol compliance is not compromised in the investigator's opinion.
4. Pregnancy or nursing, and in women of childbearing age, if they do not agree to use throughout the study a barrier contraceptive method of proven reliability in the investigator's opinion.
5. In the opinion of the principal investigator, patient is unlikely to comply with the study protocol, or the patient was not eligible for any other reason.
6. Subjects infected by the hepatitis B virus and who are being treated with tenofovir (TDF) or lamivudine (3TC).
7. Prior treatment with interferon (pegylated or not) and/or ribavirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-02; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Assess efficacy of concomitant treatment with lopinavir/r monotherapy and PEG-INF plus RBV for the control of both HIV and HCV infection respectively after 12 months of active treatment for HCV | 80 weeks

SECONDARY OUTCOMES:
Tolerability and safety of concomitant treatment with LPV/r, PEG-INF and RBV | 80 weeks
CD4 | 80 weeks
Efficacy | 80 weeks
Adherence | 80 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Ortega, Study Chair — Hospital General Universitario de Valencia
Locations (10):
- Spain (10):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Castellón, Castellon, Castellón
  - Hospital Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital General Sta. Mª del Rosell, Cartagena, Murcia
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital la Paz, Madrid
  - Hospital La Princesa, Madrid
  - Hospital La Fe, Valencia
  - Hospital General Universitario de Valencia, Valencia